CLINICAL TRIAL: NCT07150234
Title: Effectiveness of Acupuncture for Cervical Spondylotic Radiculopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Xinyu Shen, Doctor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-109-KY-01
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cervical Spondylotic Radiculopathy
Keywords: cervical spondylotic radiculopathy
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Acupuncture group received 3 acupuncture treatment sessions per week (every 1 or 2 days) over 6 weeks, 18 sessionsin total. The main acupuncture points are Jingbailao (EX-HN15), Jingjiaji (EX-B2), Binao (LI14) and Ashi. And according to the symptoms, select from the following acupoints: Wangu (GB12), Shouwuli (LI13), Quchi (LI11), Hegu (LI4), Zhongzhu (TE3) and Waiguan (TE5).
  Interventions: Device: Acupuncture
- Sham acupuncture group (Sham Comparator): Sham acupuncture group received 3 sham acupuncture treatment sessions per week (every 1 or 2 days) over 6 weeks, 18 sessionsin total. The main acupuncture points are Jingbailao (EX-HN15), Jingjiaji (EX-B2), Binao (LI14) and Ashi. And according to the symptoms, select from the following acupoints: Wangu (GB12), Shouwuli (LI13), Quchi (LI11), Hegu (LI4), Zhongzhu (TE3) and Waiguan (TE5).
  Interventions: Device: sham acupuncture

INTERVENTIONS:
Device: Acupuncture — The needles will be inserted in acupoints through adhesive pads. Needles will be lifted, thrusted and twirled gently for 3 times to achieve deqi sensation and manipulated every ten minutes.
  Arms: Acupuncture group
Device: sham acupuncture — The needles will be inserted into the pad and reaching the skin. Needles will be lifted, thrusted and twirled gently for 3 times to simulate the effect of the needle tip penetrating the skin.
  Arms: Sham acupuncture group

SUMMARY:
This study will be an evaluation of the efficacy and safety of acupuncture for cervical spondylotic radiculopathy. The main questions it aims to answer are 1. Does acupuncture improve the pain intensity among patients with cervical spondylotic radiculopathy? 2. Does acupuncture treat cervical spondylotic radiculopathy safely? Researchers will compare acupuncture to sham acupuncture to see if acupuncture could improve symptoms among patients with cervical spondylotic radiculopathy. Experimental and control groups will be treated with 6 weeks of acupuncture or sham-acupuncture respectively. Patients were followed up at 1 month, 3 months, 6 months after treatment to record outcome, any disease progression, adverse events, and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18-75 years old;
2. Patients meets the diagnostic criteria of cervical spondylotic radiculopathy and the discomfort such as pain and numbness only radiates to one upper limb (unilateral);
3. NRS score of the average 24h arm pain/numbness in the last week was ≥4;
4. The course of disease is ≥6 weeks;
5. Patients voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

1. Those with tumors, connective tissue diseases, rheumatism, spinal cord diseases, fractures, vertebral dislocation, metabolic and endocrine diseases (paget's disease, osteoporosis), other neuropathy (peripheral neuropathy, amyotrophic lateral sclerosis, transverse myelitis, Guillain-Barre syndrome, brachial plexus neuropathy), vascular related diseases (carotid artery dysfunction, arteriovenous fistula or deformity), inflammation(rheumatoid arthritis, inflammatory arthritis, ankylosing spondylitis) and infectious diseases (osteomyelitis, abscess, discitis, Lyme disease, herpes zoster, meningitis), etc.
2. Those with diseases such as scapulohumeral periarthritis, thoracic outlet syndrome, tennis elbow, carpal tunnel syndrome, etc. that cause upper limb pain or discomfort;
3. Those with cervical spondylotic radiculopathy whose condition is in a rapidly progressive stage;
4. Those received systematic comprehensive conservative treatment fails for three months, the conservative treatment includes physical therapy (fixation, traction, manipulation, exercise, ultrasound and infrared), drugs (ibuprofen, nonsteroidal anti-inflammatory drugs, gabapentin, pregabalin, antidepressants, etc.) and nerve block;
5. Those with ankylosis of vertebral joints;
6. Those neurological impairment (such as muscular atrophy and sensory disturbance);
7. Those with congenital abnormality of cervical vertebra;
8. Those with head and neck injuries and surgical history;
9. Those with long-term use of analgesics, muscle relaxants, hormones, or other pain more severe than neck pain;
10. Those with mental illness such as depression, anxiety, suicidal tendency, cognitive dysfunction or language disorder;
11. Those who received acupuncture treatment one week before joining the group;
12. Those who with drug dependence;
13. Those who with serious heart, liver, kidney, hematopoietic system, coagulation system, autoimmune system diseases, poorly controlled hypertension, diabetes, active infection, infectious diseases, severe malnutrition in the whole body, malignant tumor or serious diseases at the end stage;
14. Those who are pregnant or planning pregnancy, lactating and postpartum ≤12 months within one year;
15. Those who are metal allergy or serious needle fear;
16. Those with skin ulcer, damage and scar at selected acupoints;
17. Those who have received other clinical study within 90 days prior to randomization;
18. Pending litigation or industrial injury compensation related to neck pain;
19. Those who are unable to communicate in Mandarin or read Chinese.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | At 6 weeks from randomization.
  Average NRS (numerical rating scale) score of arm pain decreased by at least 30% compared with baseline in the past 24 hours.

SECONDARY OUTCOMES:
The average NRS (numerical rating scale) score of arm pain in the past 24 hours as change from baseline. | At 1,3,6,10,18,30 weeks from randomization.
The average NRS (numerical rating scale) score of neck pain in the past 24 hours as change from baseline. | At 1,3,6,10,18,30 weeks from randomization.
Clinical response rate | At 1,3,10,18,30 weeks from randomization.
  NRS (numerical rating scale) score of arm pain decreased by at least 30% compared with baseline in the past 24 hours.
Clinical response rate | At 1,3,6,10,18,30 weeks from randomization.
  NRS (numerical rating scale) score of neck pain decreased by at least 30% compared with baseline in the past 24 hours.
The NDI (Neck Disability Index) score as change from baseline. | At 3,6,10,18,30 weeks from randomization.
Percentage of patients with NDI (Neck Disability Index) score lower than baseline by 8.5 points or more. | At 3,6,10,18,30 weeks from randomization.
NRS (numerical rating scale) score of the maximum neck/arm pain during neck exercise as change from baseline. | At 1,3,6,10,18,30 week from randomization.
ISI-C (Insomnia Severity Index) score as change from baseline. | At 6,10,18,30 weeks from randomization.
PHQ-9 (Patient Health Questionnaire-9) score as change from baseline. | At 3,6,10,18,30 weeks from randomization.
GAD-7 (Generalized Anxiety Disorder-7) score as change from baseline. | At 3,6,10,18,30 weeks from randomization.
EQ-5D-5L score as change from baseline. | At 6,10,18,30 weeks from randomization.
Patient Global Impression of Change, PGIC | At 6,30 weeks from randomization.
  1 means great improvement of arm pain, 2 means moderate improvement of arm pain, 3 means better of arm pain, 4 means no change of arm pain, 5 means slight deterioration of arm pain, 6 means moderate deterioration of arm pain and 7 means much deterioration of arm pain.
Percentage of emergency painkillers used in the past week. | At 1,3,6,10,18,30 weeks from randomization.
The total number of days of using emergency painkillers in the past week. | At 1,3,6,10,18,30 weeks from randomization.
Adverse event | At 1,3,6,10,18,30 weeks from randomization.
  Collect the adverse reactions related to acupuncture, such as needle breakage, local hematoma, infection and abscess, and any unexpected symptoms, signs or health conditions during the experiment.

OTHER OUTCOMES:
Assessment of belief in acupuncture | Baseline assessment (week 0)
  Participants will be asked: Do you think your cervical spondylotic radiculopathy may be helped by acupuncture?
Blinding assessment Description | Within 5 minutes after either treatment at week 6.
  Participants will be asked: Do you think you have received traditional acupuncture in the past 6 weeks?

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with the publication until six months after publication.
Access Criteria: A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal.